CLINICAL TRIAL: NCT01528488
Title: A Randomized, Double-blind, Prospective Trial of Prophylactic EVOZAC® Calming Skin Spray for EGFR-TKIs Associated Rash Eruption in Non-small Cell Lung Cancer
Brief Title: Prophylactic EVOZAC® Calming Skin Spray for EGFR-TKIs Associated Rash Eruption in NSCLC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EVOZAC20110210
Record Dates: First submitted 2012-02-03; First posted 2012-02-08 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EVOZAC (Experimental): EVOZAC should be sprayed to the skin of the total face three times per day.
  Interventions: Other: EVOZAC Calming Skin Spray
- Physiological saline (Placebo Comparator): Physiological saline should be sprayed to the total face three times per day.
  Interventions: Other: Physiological saline

INTERVENTIONS:
Other: EVOZAC Calming Skin Spray — EVOZAC Calming Skin Spray should be sprayed to the skin in the total face, three times per day
  Arms: EVOZAC
Other: Physiological saline — Physiological saline was used as the placebo of EVOZAC® Calming Skin Spray and should be also sprayed on the total face, three times per day
  Arms: Physiological saline

SUMMARY:
The epidermal growth factor receptor (EGFR) has become an important target for cancer therapy, and the small molecular tyrosine kinase inhibitors (EGFR-TKIs) have played an important role in the treatment of non-small cell lung cancer (NSCLC). What accompanies with the encouraging efficacy in NSCLC is the common side effects, of which the most common one is the specific papular and pustular acne-like rash which affects mainly the face, scalp, and upper torso. But till now, no medicament has been proved effective enough to treat or prevent the EGFR-TKIs associated rash. The EVOZAC® Calming Skin Spray has shown acceptable activity at the rash prevention in our preliminary study, so the investigators conduct the randomized, double-blind, controlled trial to evaluate the efficacy and safety of EVOZAC® Calming Skin Spray in prevention of EGFR-TKIs associated rash in NSCLC.

DETAILED DESCRIPTION:
Not suitable: no more information is needed to be described.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven NSCLC diagnosis
* Life expectancy over four weeks
* absolute neutrophil count ≥ 2.0X109/L, Pt ≥ 100X109/L, hemoglobin ≥ 90g/l
* With normal hepatic function(AST, ALT < 2.5 x upper limit of normal , and Total bilirubin ≤ upper limit of normal)
* Suitable for EGFR-TKIs treatment and expectant duration over four weeks
* No specific therapies received within 4 weeks prior to enrollment which may induce similar skin reaction,such as Cetuximab, Sorafenib, Avastin.
* With a pre-existing peripheral neuropathy (National Cancer Institute Common Toxicity Criteria for Adverse Events [NCI-CTC] grade ≥ 3)
* No other concomitant therapy referred to the face skin during the study
* Signed and dated informed consent

Exclusion Criteria:

* Performance status ≥ 3(ECOG)
* Pregnant or breast-feeding patients
* The lesion counts can't be evaluated due to concomitant diseases or other conditions
* Not suitable for EGFR-TKIs treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Lesion counts in total face at completion of the study period (week 4) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: li zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Medical Oncology,Cancer Center of Sun Yat-Sen University, Guangzhou, Guangdong, China